CLINICAL TRIAL: NCT06041204
Title: Letrozole Alone vs. Letrozole Plus Levothyroxine for Ovulation Induction in Infertile Women With Both (Polycystic Ovary Syndrome) PCOS and Sub-clinical Hypothyroidism.
Brief Title: Best Treatment for Women With Both (Polycystic Ovary Syndrome) PCOS and Subclinical Hypothyroidism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy (Other)
Responsible Party: Sponsor-Investigator, Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy, lecturer and consultant at Obstetrics and Gynecology Department., Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gyne2021
Record Dates: First submitted 2023-09-05; First posted 2023-09-18 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries; Subclinical Hypothyroidism; Female Infertility
Keywords: Letrozole; Levothyroxine; PCOS; Subclinical hypothyroidism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility, Female | interventions — Letrozole; Thyroxine; Tablets

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letrozole Group (Active Comparator): Participants randomized to letrozole group will take 5mg tablets orally daily for 5 days starting on day 3 of cycle. Dose can be adjusted up to 7.5mg based on ovulation response, maintained for subsequent cycles. Treatment continues for up to 6 ovulatory cycles or until pregnancy occurs. Ovulation assessed by follicular monitoring and progesterone. Compliance monitored by pill counts and diary. Routine antenatal care if pregnant. Adverse effects monitored per guidelines. Participants followed for multiple pregnancies. Tablets taken at same time each day. Maximum treatment period is 6 months.
  Interventions: Drug: Letrozole 2.5mg
- Letrozole plus levothyroxine (Experimental): Participants randomized to this group will take letrozole tablets at same dose and schedule as letrozole only group. In addition, they will take levothyroxine tablets orally once daily. Levothyroxine dose will start at 25mcg and be titrated based on TSH level, with a target TSH in the normal range. Participants will take levothyroxine at approximately same time each day. Letrozole dosing and schedule as described for other group. Treatment continues for up to 6 ovulatory cycles or until pregnancy occurs. Ovulation assessed by follicular monitoring and progesterone. Compliance monitored by pill counts, TSH levels and diary. Routine antenatal care if pregnant. Adverse effects monitored per guidelines. Participants followed for multiple pregnancies. Maximum treatment period is 6 months.
  Interventions: Drug: Letrozole 2.5mg; Drug: Levothyroxine 25 Mcg (0.025 Mg) Oral Tablet

INTERVENTIONS:
Drug: Letrozole 2.5mg — Participants will receive 2.5mg letrozole tablets orally daily for 5 days starting on day 3 of menstrual cycle. The 2.5mg dose will be maintained for at least the first 3 cycles. If no ovulation after 3 cycles, dose cautiously increased up to 7.5mg maximum. Once minimum ovulation dose determined, it will be continued for up to 6 cycles total or until pregnancy occurs. Compliance monitored by pill counts and diary. Ovulation assessed by follicular monitoring and progesterone levels. Routine antenatal care if pregnant. Adverse effects monitored and managed per guidelines. Participants followed for multiple pregnancies. Maximum treatment duration is 6 ovulatory cycles or 6 months. Tablets taken at same time each day.
Drug: Levothyroxine 25 Mcg (0.025 Mg) Oral Tablet — Participants will take letrozole at same doses as letrozole only group. Also receive levothyroxine starting at 25mcg orally once daily, titrated by 25mcg every 4 weeks to reach normal TSH, maximum 100mcg daily. Once appropriate dose determined to normalize TSH, it is maintained throughout treatment period. Compliance monitored by pill counts, TSH levels, and diary. Treatment continues for up to 6 ovulatory cycles or until pregnancy, whichever is first, maximum 6 months. Ovulation assessed by monitoring and progesterone. Routine antenatal care if pregnant. Adverse effects monitored and managed per guidelines. Participants followed for multiple pregnancies. Letrozole and levothyroxine taken daily at same time. All other procedures same as letrozole only group.
  Other Names: levothyroxine 25
  Arms: Letrozole plus levothyroxine

SUMMARY:
The goal of this randomized controlled trial is to compare letrozole alone versus letrozole plus levothyroxine for ovulation induction in infertile women with both PCOS and subclinical hypothyroidism. The main questions it aims to answer are:

Is letrozole plus levothyroxine superior to letrozole alone in achieving ovulation in these patients? Does combining levothyroxine with letrozole lead to higher pregnancy and live birth rates compared to letrozole alone?

Participants will be randomized into two groups:

Group 1 will receive letrozole only, starting at 2.5 mg daily from day 3 to 7 of the menstrual cycle. The dose will be increased up to 7.5 mg if no ovulation occurs, for a maximum treatment period of 6 months or until pregnancy is achieved.

Group 2 will receive letrozole at the same doses as group 1 plus 25 mcg levothyroxine daily.

ELIGIBILITY:
Inclusion Criteria:

Age between 20-40 years

BMI between 18-35 kg/m2

Meet diagnostic criteria for PCOS based on the Rotterdam consensus criteria and ESHRE/ASRM modifications (2018):

Oligo- and/or anovulation Clinical and/or biochemical signs of hyperandrogenism Polycystic ovaries on ultrasound

Subclinical hypothyroidism defined as TSH level between 5-10 mIU/L with normal free T4

Infertility duration ≥ 1 year

Intact ovaries and uterus, confirmed by physical exam and imaging

Normal semen analysis in male partner

No tubal or peritoneal factor contributing to infertility

Effective contraception if not attempting conception

Willing and able to provide informed consent

Exclusion Criteria:

Known thyroid disease or on thyroid medications

Abnormal thyroid function tests other than subclinical hypothyroidism

Hyperprolactinemia

Presence of other causes of infertility such as:

Moderate to severe male factor infertility Bilateral tubal occlusion or peritoneal factors Stage III-IV endometriosis Ovarian failure or insufficiency (high FSH or low AMH)

Previous diagnosis of any type of congenital adrenal hyperplasia

Uncontrolled diabetes (HbA1C >8%)

History of deep vein thrombosis or thromboembolic events

Any contraindication to letrozole or levothyroxine

Previous use of letrozole or levothyroxine in past 6 months

Current or suspected pregnancy

Breastfeeding

Inability to comply with treatment and follow-up procedures

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study will only enroll female participants. Patients must be of reproductive age with intact uteri and ovaries to meet the inclusion criteria.
  The study aims to induce ovulation for conception in infertile women with PCOS and subclinical hypothyroidism. As such, only individuals biologically born as females and currently identifying as women will be eligible.
  All enrolled participants must have functioning ovaries and intact reproductive organs capable of sustaining a pregnancy. Patients who have undergone surgical sterilization procedures like tubal ligation or hysterectomy will be excluded.
  Confirmation of female gender will be through medical history, physical examination, and review of medical records if needed. Pregnancy tests will be done at screening and before each treatment cycle.
  The reproductive status, ovaries and uterus will be assessed by medical history, physical examination and imaging like ultrasound when indicated.
Enrollment: 200 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | Assessed at the end of each cycle. the cycles are 6. Each cycle is 28 days.
  Biochemical evidence of pregnancy by positive urine or serum β-hCG test.
Live birth rate | Through study completion average 1 year.
  The number of deliveries that resulted in a live born baby, documented by hospital delivery records.

SECONDARY OUTCOMES:
Ovulation rate | Assessed at the end of each cycle. the cycles are 6. Each cycle is 28 days.
  Evidence of ovulation by ultrasound monitoring of dominant follicle development and serum progesterone level > 3 ng/mL in mid-luteal phase.
Miscarriage rate | Through study completion average 1 year.
  Loss of clinical pregnancy before 20 weeks gestation, confirmed by ultrasound or histopathology.
Menstrual regularity | Through study completion average 1 year.
  Normal ovulatory menstrual cycles defined as cycle length 21-35 days.
Side effects | Through study completion average 1 year.
  Participant reports of adverse effects of letrozole or levothyroxine, graded per standard criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Muhamed Alhagrasy, M.D., Principal Investigator — Al-Azhar University
Locations (1):
- Al-Hussein University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
To protect participant confidentiality, individual-level data from this study will not be made publicly available. However, de-identified aggregated data and results can be shared with other researchers upon request after publication. Any data provided will be limited, non-identifiable, and subject to a data use agreement to ensure participant privacy. Only select excerpts needed to validate findings will be shared under approved research objectives. The investigators reserve the right to reject requests that may compromise anonymity. We aim to promote transparency through controlled data access rather than public availability of the full dataset due to re-identification risks for participants.